CLINICAL TRIAL: NCT03293472
Title: Inflammatory Mediators, Neural Tissue Injury Markers and the Markers of Oxidative Stress in the CSF of Patients Undergoing Spinal Anesthesia With Ropivacaine and Bupivacaine
Brief Title: Neurotoxicity of Spinal Anesthesia With Ropivacaine and Bupivacaine
Acronym: BuRoNe
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rzeszow (Other)
Collaborators: Department of Anesthesiology, Intensive Therapy, District Hospital No2 in Rzeszow (Unknown)
Responsible Party: Principal Investigator, Marek Wojtaszek, M.D., Ph.D., University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URzeszow
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural; Anaesthetic Complication Neurological
MeSH Terms: interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Parallel study
Who Masked: Participant
Masking Description: Patient unaware of the local anesthetic used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Experimental): Experimental: 0.5% ropivacaine (isobaric) 4.5 ml for the patients < 160 cm tall, 5.0 ml for 161-170 cm tall, 5.5 ml for 171-180 cm tall, and 6.0 ml > 180 cm.
  supplementary bolus doses of ropivacaine as required, followed by 0.2% ropivacaine, 1 ml/h for the postoperative period
  Interventions: Drug: Ropivacaine
- Bupivacaine (Active Comparator): 0.5% v Bupivacaine mg (isobaric) loading dose of 0.5% bupivacaine, 3.0 ml for the patients < 160 cm tall, 3.3 ml for 161-170 cm tall, 3.6 ml for 171-180 cm tall, and 4.0 ml > 180 cm.
  and supplementary bupivacaine bolus dose as required, followed by 0,12% bupivacaine 1 ml/h for the postoperative period
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Ropivacaine — Procedure: Continuous Epidural Anesthesia Local anesthetic injection to the cerebrospinal fluid (subarachnoid space) at the L3-L4 or L4-L5 level Drug: ropivacaine Other name: Ropimol 0.5% ropivacaine (isobaric) 4.5 ml for the patients < 160 cm tall, 5.0 ml for 161-170 cm tall, 5.5 ml for 171-180 cm tall, and 6.0 ml > 180 cm, supplementary ropivacaine bolus doses as required, followed by 0.2% ropivacaine, 1 ml/h for the postoperative period Device : The Wiley Spinal Catheter-Over-Needle System for Continuous Spinal Anesthesia 4-6" 23-gauge intrathecal cannula over a 27-gauge pencil-point spinal needle
  Other Names: Ropimol
  Arms: Ropivacaine
Drug: Bupivacaine — Procedure: Continuous Epidural Anesthesia Local anesthetic injection to the subarachnoid space at the L3-L4 or L4-L5 level Drug: bupivacaine Loading dose of bupivacaine followed by 0.12% bupivacaine, 1 ml/h Other name: bupivacaine
  Device:
  The Wiley Spinal Catheter-Over-Needle System for Continuous Spinal Anesthesia 4-6" 23-gauge intrathecal cannula over a 27-gauge pencil-point spinal needle
  Arms: Bupivacaine

SUMMARY:
Consenting patients, scheduled for orthopaedic surgery under spinal anesthesia will be randomly assigned (1:1) to receive ropivacaine or bupivacaine as a single shot before the start of surgery, followed by bolus doses of the same local anesthetic as required during the surgery, and continuous infusion of the same local anesthetic for 24 hours postoperatively.

Primary Outcome Measures: Evaluation of changes in concentrations of glutamate in the cerebrospinal fluid and in the blood. Secondary outcomes: : Evaluation of changes in concentrations of selected mediators of inflammatory response (IL-1β, IL-6, TNF and others) and selected chemokines as markers of the glia damage.

Hemodynamic stability during the surgery, and efficacy of postoperative analgesia will be also evaluated.

DETAILED DESCRIPTION:
With the approval from the Bioethical Committee of the University of Rzeszow, informed written consent will be obtained from all patients.

A sample size of 60 patients was calculated to obtain at least 25% reduction of glutamate concentration in the cerebrospinal fluid in the ropivacaine group with 0,05 significance and power of 0,8.

Consenting patients, scheduled for orthopaedic surgery under spinal anesthesia will be randomly (1:1) assigned using closed envelopes to receive intrathecally ropivacaine or bupivacaine as a single shot before the start of surgery, followed by bolus doses of the same local anesthetic as required during the surgery, and continuous infusion of the same local anesthetic for 24 h for postoperative pain relief. All block will be performed in the sitting position, and the drug will be administered in supine position through the catheter in the intrathecal space. Blood and cerebrospinal fluid samples will be drawn at predetermined time intervals centrifuged as required and frosen in -70deg C until analysis.

Eligibility Ages eligible for study 18 years and older (Adult, Senior) Sexes Eligible for the Study: All Accepts Healthy Volunteers: No

Inclusion Criteria:

Orthopedic procedures in the lower limbs Written informed consent Exclusion criteria Patients' refusal Known allergies to study medications Anatomic, posttraumatic and postoperative deformations of the spinal column making placement of intrathecal catheter impossible Neurological contraindications Any other contraindications for spinal anesthesia (coagulations disorders, antiplatelet or anticoagulant treatment, infection at the puncture site.

Inability to comprehend or participate in pain scoring scale

ELIGIBILITY:
Inclusion Criteria:

- Orthopedic procedures in the lower limbs Written informed consent

Exclusion Criteria:

* Patients' refusal Known allergies to study medications Inability to comprehend or participate in pain scoring scale Anatomic, posttraumatic and postoperative deformations of the spinal column making placement of intrathecal catheter impossible Neurological contraindications Any other contraindications for spinal anesthesia (coagulations disorders, antiplatelet or anticoagulant treatment, infection at the puncture site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory mediators, neural tissue injury markers and the markers of oxidative stress in the cerebrospinal fluid of patients undergoing spinal anesthesia with ropivacaine and bupivacaine. | 24 h
  Evaluation of changes in concentrations of
  • glutamate in the cerebrospinal fluid and in the blood of patients undergoing orthopaedic surgery under spinal anesthesia with either ropivacaine or bupivacaine

SECONDARY OUTCOMES:
Inflammatory mediators, neural tissue injury markers and the markers of oxidative stress in the cerebrospinal fluid of patients undergoing spinal anesthesia with ropivacaine and bupivacaine. | 24 h
  Evaluation of changes in concentrations of selected mediators of inflammatory response (IL-1β, IL-6, tumor necrosis factor and others)
Inflammatory mediators, neural tissue injury markers and the markers of oxidative stress in the cerebrospinal fluid of patients undergoing spinal anesthesia with ropivacaine and bupivacaine. | 24 h
  Evaluation of changes in concentrations of • selected chemokines as markers of the glia damage in the cerebrospinal fluid and in the blood of patients undergoing orthopaedic surgery under continuous spinal anesthesia with either ropivacaine or bupivacaine

OTHER OUTCOMES:
Inflammatory mediators, neural tissue injury markers and the markers of oxidative stress in the CSF of patients undergoing spinal anesthesia with ropivacaine and bupivacaine. | 24 h
  Assessment of hemodynamic stability in patients anaesthetized with continuous epidural infusion of ropivacaine and bupivacaine
Inflammatory mediators, neural tissue injury markers and the markers of oxidative stress in the CSF of patients undergoing spinal anesthesia with ropivacaine and bupivacaine. | 24h
  Postoperative pain severity in Numerical Rating Scale (NRS) in the first 24 hours after surgery [Time Frame: 24 h] NRS range from 0 for no pain to 10 for worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszow, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wille M. Intrathecal use of ropivacaine: a review. Acta Anaesthesiol Belg. 2004;55(3):251-9. PMID 15515303
- [Result] Kuthiala G, Chaudhary G. Ropivacaine: A review of its pharmacology and clinical use. Indian J Anaesth. 2011 Mar;55(2):104-10. doi: 10.4103/0019-5049.79875. PMID 21712863
- [Result] Sung CM, Hah YS, Kim JS, Nam JB, Kim RJ, Lee SJ, Park HB. Cytotoxic effects of ropivacaine, bupivacaine, and lidocaine on rotator cuff tenofibroblasts. Am J Sports Med. 2014 Dec;42(12):2888-96. doi: 10.1177/0363546514550991. Epub 2014 Oct 8. PMID 25296645